CLINICAL TRIAL: NCT02686281
Title: A Double-Blind, Placebo-Controlled, Randomised, Two Part Study of the Safety and Pharmacokinetics of GMC-252 in A) Healthy Male Subjects, Including a Comparison of GMC-252 Dosing in the Fed and Fasted States ,and B) in Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Pharmacokinetics Study of a New Drug for Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reason
Sponsor: Genmedica Therapeutics S.L. (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GMC-252-1.02
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Part A) (Experimental): Single ascending oral administrations of GMC-252-L-Lysine Salt and matching placebo
  Interventions:
  Drug: GMC-252-L-Lysine Other: Placebo
  Interventions: Drug: GMC-252-L-Lysine; Other: Placebo
- Cohort B (Part A) (Experimental): Single ascending oral administrations of GMC-252-L-Lysine Salt and matching placebo
  Interventions:
  Drug: GMC-252-L-Lysine Other: Placebo
  The dose administered in Part A (fed) was based on the outcome of Part A (fasted).
  Interventions: Drug: GMC-252-L-Lysine; Other: Placebo

INTERVENTIONS:
Drug: GMC-252-L-Lysine
Other: Placebo

SUMMARY:
The purpose of this study is to determine the toxicity, tolerability and safety of single ascending doses of GMC-252-L-Lysine Salt in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) within the range of 18-35 kg/m2 inclusive. BMI = Body weight (kg) / [Height (m)]2.
* Diet: Able to eat standard food, no vegetarians.
* Compliance: Understood and was willing, able and likely to comply with all study procedures and restrictions.
* Consent: Demonstrated understanding of the study and willingness to participate as evidenced by voluntary written informed consent and had received a signed and dated copy of the Informed Consent Form.
* Had no known hypersensitivity to diflunisal, NAC (N-acetylcysteine) or other non-steroidal anti-inflammatory drugs (NSAIDs).
* Had no known peptic ulcer diseases.
* Had an estimated creatinine (CREA) clearance ≥ 50 mL/min (Creatinine clearance was calculated from the serum CREA value using the Cockroft & Gault formula).
* Had no history of heart failure or uncontrolled hypertension or other known overt cardiovascular disease.
* Had no history of 'Aspirin Triad' (chronic rhinosinusitis with polyps, severe asthma and intolerance to aspirin or other NSAIDs).
* Had no marked abnormality of liver tests before entry into the study.
* Male subject willing to use an effective method of contraception, if applicable (unless anatomically sterile or where abstaining from sexual intercourse was in line with the preferred and usual lifestyle of the subject) from Day 1 until 3 months afterwards.
* Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values at the Screening Visit.
* Subject with a negative urinary drugs of abuse screen (a positive alcohol result could have been repeated at the discretion of the Investigator).
* Subject with negative human immunodeficiency virus (HIV) and Hepatitis B (Hep B) and Hepatitis C (Hep C) results.
* Subject with no clinically significant abnormalities in 12-lead ECG at the Screening Visit.
* Subject was available to complete the study (including all Follow-up Visits).
* Subject satisfied a medical examiner about their fitness to participate in the study.
* Subjects were non-smokers and non-alcohol drinkers or drank alcohol in moderation (e.g. ≤ 14 units/week).

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
* Receipt of regular medication at the Screening Visit that may have had an impact on the safety and objectives of the study (at the Investigator's discretion).
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* A clinically significant history of previous allergy/sensitivity to GMC-252.
* A clinically significant history of drug or alcohol abuse.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 16 weeks or a marketed drug clinical study within the previous 12 weeks. (N.B. washout period between trials defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
* Donation of 450 mL or more blood within the previous 12 weeks.
* Receipt of any medication since the Screening Visit that may have had an impact on the safety and objectives of the study (at the Investigator's discretion).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Over a 14 days period post dose
  Physical status (Vital signs; 12-lead ECG; Urinalysis; Haematology and biochemistry)

SECONDARY OUTCOMES:
Maximal Concentration (Cmax) | Over a 14 days period post dose
Area Under the Concentration-Time Curve | Over a 14 days period post dose

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, MBBS, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided